CLINICAL TRIAL: NCT04990999
Title: Vestibular Extraction Technique (VET): a Novel Atraumatic Extraction Technique (Randomized Clinical Trial)
Brief Title: Vestibular Extraction Technique (VET): a Novel Atraumatic Extraction Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: vestibular extraction 2021
Record Dates: First submitted 2021-07-26; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Tooth Extraction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vestibular Root Extraction (Experimental)
  Interventions: Procedure: Vestibular Root Extraction
- Atraumatic extractions using periotomes followed by conventional forceps (Active Comparator)
  Interventions: Procedure: Atraumatic extractions using periotomes followed by conventional forceps

INTERVENTIONS:
Procedure: Vestibular Root Extraction — a 1-cm long vestibular access incision was cut, 3-4 mm apical to the mucogingival junction of the involved tooth, then pushing the vestibular pouch in an incisal direction exposing the apical root area, and allowing direct undisturbed access to the root surface
  Arms: Vestibular Root Extraction
Procedure: Atraumatic extractions using periotomes followed by conventional forceps — a sulcular releasing incision suing a micro scalpel was made to detach the surrounding tissues, followed by applying the periotome interproximally into the PDL space, widening the attached periodontal ligaments space.
  Arms: Atraumatic extractions using periotomes followed by conventional forceps

SUMMARY:
study proposes an alternative atraumatic tooth extraction procedure; Apically achieved exodontia, which might offer an alternative to the conventional incisal exodontia, whilst providing minimum tissue trauma and subsequently maximum marginal tissue preservation.

DETAILED DESCRIPTION:
A sample of 26 patients that received the extraction therapy For Group (A) patients, Atraumatic extractions using periotomes followed by conventional forceps were performed.

For Group (B) patients, the novel technique of Vestibular Root Extraction was performed to the sample group's hopeless teeth.

ELIGIBILITY:
Inclusion Criteria:

* Single non-adjacent hopeless maxillary anterior teeth
* Type II socket)
* Intact overlying soft tissues.
* Adequate palatal and at least 3 mm apical bone

Exclusion Criteria:

* Smokers
* Pregnant females
* Patients with systemic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Changes in post restorative soft tissue height | at baseline and 12 months
  identified midfacially and at the apex of the mesial and distal papillae by superimposing the STL (Standard Triangle Language) files of the models, obtained via IOS

CONTACTS AND LOCATIONS:
Locations (1):
- Private Practice Clinic, Alexandria, Egypt